CLINICAL TRIAL: NCT03773068
Title: Open Label, Partially Randomized, Cross-over Study to Determine the Absolute Bioavailability and Pharmacokinetics of BAY1817080 Using a Simultaneous Anticipated Therapeutic Oral Dose Along With an i.v. [13C715N]-Labeled Microtracer and to Investigate the Relative Bioavailability of Two Formulations Given Under Different Diets at 2 Dose Levels in Healthy Volunteers
Brief Title: A Study in Healthy Volunteers Investigating How Quickly and to What Extent BAY1817080 is Taken up, Distributed, Broken Down and Eliminated From the Body, as Well as the Difference Between 2 Different Types of Tablets of BAY1817080 and the Difference Between Oral Dose and Dose in the Vein
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 19519; 2018-001814-13 (EudraCT Number)
Record Dates: First submitted 2018-12-04; First posted 2018-12-12 (Actual); Last update posted 2019-08-19 (Actual); Status verified 2019-08

CONDITIONS: Biological Availability
Keywords: Endometriosis; Refractory chronic cough
MeSH Terms: conditions — Endometriosis; Chronic Cough

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Group 1 - BAY1817080 Dose 1 (Experimental): Participants will receive one single oral dose of BAY1817080 - Formulation B at dose 1 under fasted condition
  Interventions: Drug: BAY1817080 - Formulation B
- Group 2 - BAY1817080 Dose 2 (Experimental): Participants will receive a) one single oral dose of BAY1817080 - Formulation A at dose 2 with moderate-fat, moderate-calorie meal (MF, MC); b) one single oral dose of BAY1817080 - Formulation B at dose 2 along with one intravenous (i.v.) infusion of 0.1 mg [13C715N]-BAY1817080; and c) one single oral dose of BAY1817080 - Formulation B at dose 2 with high-fat, high-calorie meal (HF, HC). The 3 treatments will be administered with a randomized sequence
  Interventions: Drug: BAY1817080 - Formulation A; Drug: BAY1817080 - Formulation B; Drug: [13C715N]-BAY 181708 stable isotope label (SIL)
- Group 3 - BAY1817080 Dose 3 (Experimental): Participants will receive a) one single oral dose of BAY1817080 - Formulation B at dose 3 under fasted condition; followed by one single oral dose of BAY1817080 - Formulation A at dose 3 with MF, MC; and followed by one single oral dose of BAY1817080 - Formulation B at dose 3 with HF, HC. The 3 treatments will be administered with a fixed sequence
  Interventions: Drug: BAY1817080 - Formulation A; Drug: BAY1817080 - Formulation B

INTERVENTIONS:
Drug: BAY1817080 - Formulation A — Formulation A
  Arms: Group 2 - BAY1817080 Dose 2; Group 3 - BAY1817080 Dose 3
Drug: BAY1817080 - Formulation B — Formulation B
Drug: [13C715N]-BAY 181708 stable isotope label (SIL) — 0.1 mg [13C715N]-BAY181708, 15 minutes i.v. infusion at the estimated tmax after administration of Formulation B
  Arms: Group 2 - BAY1817080 Dose 2

SUMMARY:
The main purpose of this study is to investigate how quickly and to what extent BAY1817080 is absorbed (taken up), distributed, metabolized (broken down) and eliminated from the body (this is called pharmacokinetics). The pharmacokinetics of BAY1817080 administered as tablets will be compared to the pharmacokinetics of BAY1817080 administered as intravenous (iv; in the vein) infusion (this is called absolute bioavailability). Furthermore, 2 different types of tablets with BAY1817080 (Formulation A and Formulation B) will be compared with regard to pharmacokinetics (this is called relative bioavailability). The effect of a meal on the pharmacokinetics of BAY1817080 administered as tablets will be investigated as well. Finally, it will also be investigated how safe BAY1817080 is and how well BAY1817080 is tolerated.

ELIGIBILITY:
Inclusion criteria:

* Healthy male subject
* Age: 18 to 55 years (inclusive) at the time of informed consent and first dose of study medication
* Body mass index (BMI) above/equal to 18 and below/equal to 30 kg/m^2 at Screening
* Body weight of at least 45 kg at Screening

Exclusion criteria:

* Presence or history of clinically relevant cardiovascular, central nervous system (CNS), hepatic, hematopoietic disease, renal dysfunction, metabolic or endocrine dysfunction, serious allergy, asthma hypoxemia, hypertension, seizures, or allergic skin rash
* Known hypersensitivity to the study drugs
* Known severe allergies or significant non-allergic drug reactions
* Febrile illness within 1 week before study drug administration
* Current or recent (within 6 months) gastrointestinal disease that would be expected to influence the absorption of drugs
* Subject has a history of cancer, except basal cell carcinoma which has been in remission for at least 5 years prior to Screening
* Poor peripheral venous access
* Regular use of medicines within 6 months prior to screening
* Clinically relevant findings in the electrocardiogram (ECG), physical examination or laboratory examination

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2018-12-13 (Actual); Primary Completion 2019-06-21 (Actual); Study Completion 2019-08-12 (Actual)

PRIMARY OUTCOMES:
Absolute oral bioavailability (F) of BAY1817080 | Up to 10 days
Relative bioavailability (frel) of Formulation A versus Formulation B given under different diets | Up to 10 days

SECONDARY OUTCOMES:
Effect of a high-fat, high-calorie meal (HF,HC) on the PK of BAY1817080 after a single oral dose of Formulation B at two doses in comparison to the fasted state evaluated by Cmax | Up to 10 days
  Maximum observed drug concentration in plasma after single dose administration (Cmax) of BAY1817080 will be analyzed assuming log-normally distributed data.
Effect of a high-fat, high-calorie meal (HF,HC) on the PK of BAY1817080 after a single oral dose of Formulation B at two doses in comparison to the fasted state evaluated by AUC | Up to 10 days
  Area under the concentration versus time curve from zero to infinity after single dose administration (AUC) of BAY1817080 will be analyzed assuming log-normally distributed data. AUC from time 0 to the last data point greater than lower limit of quantification (AUC[0-tlast]) will be used if AUC cannot be calculated reliably in all subjects.
Dose proportionality in BAY1817080 PK after a single oral dose of Formulation B across three doses in fasted state evaluated by Cmax/D | Up to 10 days
  To investigate dose-proportionality, Cmax divided by dose (Cmax/D) derived from the 3 oral doses of Formulation B in fasted state will be analyzed.
Dose proportionality in BAY1817080 PK after a single oral dose of Formulation B across three doses in fasted state evaluated by AUC/D | Up to 10 days
  To investigate dose-proportionality, AUC divided by dose (AUC/D) derived from the 3 oral doses of Formulation B in fasted state will be analyzed. AUC(0-tlast)/D will be used if AUC/D cannot be calculated reliably in all subjects.
Frequency and severity of treatment emergent adverse events (TEAEs) | Up to 42 days

CONTACTS AND LOCATIONS:
Locations (1):
- PRAHealthSciences, Groningen, Netherlands

REFERENCES:
- [Derived] Francke K, Chattopadhyay N, Klein S, Rottmann A, Krickau D, van de Wetering J, Friedrich C. Preclinical and Clinical Pharmacokinetics and Bioavailability in Healthy Volunteers of a Novel Formulation of the Selective P2X3 Receptor Antagonist Eliapixant. Eur J Drug Metab Pharmacokinet. 2023 Jan;48(1):75-87. doi: 10.1007/s13318-022-00805-5. Epub 2022 Dec 5. PMID 36469250